CLINICAL TRIAL: NCT04154085
Title: Narrative Therapy for Treatment-Resistant Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Justine Dembo, Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4136016
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Narrative therapy; Group therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: A group consisting of 12-15 participants will be recruited for this initial exploratory study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): This study only has one arm; all patients receive the treatment intervention.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — Group psychotherapy

SUMMARY:
This is a prospective exploratory study using narrative therapy in group format, over 20 sessions, 2 hours per session, weekly, to determine whether this modality can provide any benefit to OCD symptoms, mood, sense of social connectedness, sense of identity, and/or quality of life in individuals living with treatment-resistant OCD. NOTE: an amendment is now in place so that the group can occur virtually given the COVID pandemic; Zoom will be used as our platform.

DETAILED DESCRIPTION:
Many patients referred to the Thompson Centre at Sunnybrook have severe OCD, and have significant and disabling symptoms even after completing our treatment protocols, including our intensive and residential programs. These patients have already undergone traditional cognitive behavioural therapy (CBT) and exposure and response prevention (ERP), as well as pharmacotherapy. Patients voice distress at their poor quality of life and high symptom burden, and can feel hopeless, if they have exhausted numerous evidence-based treatment options without significant improvement. Narrative therapy is a unique approach, based on the premise that language reflects a social construction of reality. Individuals with severe mental illness hold within themselves life narratives that reinforce their painful beliefs about themselves, the world, and others. Evidence indicates that narrative therapy can help to create a more cohesive identity and a more flexible view of the self and the future.

Our primary goal is to determine whether narrative therapy could improve OCD symptom burden and quality of life in a highly treatment-resistant population. Domains such as mood, identity, and interpersonal connectedness are secondary measures. The research questions are: could narrative therapy lead to symptomatic improvement in treatment-resistant OCD? And could narrative therapy improve the domains of mood, interpersonal connectedness, and/or identity in patients with treatment-resistant OCD?

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and write fluently in English.
* Patients who have participated in the intensive/residential program or group programs and/or have received pharmacotherapy with a psychiatrist at the Frederick W. Thomspon Anxiety Disorder Centre
* Patients between the ages of 18-65
* Only patients who have treatment-resistant OCD are eligible. For the purposes of this study we are defining this as: failure to achieve remission after having tried 1) At least two first-line SSRI's AND either clomipramine or atypical antipsychotic augmentation, and 2) at least one full course of exposure and response prevention (ERP), or our intensive/residential program.

Exclusion Criteria:

* those with active substance abuse/dependence within three months
* suspected organic pathology
* recent suicide attempt/active suicidality
* current self-injurious behaviour
* active bipolar or psychotic disorder
* history of aggression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
YBOCS Change | Prior to start; at 5 weeks, 10 weeks, 15 weeks, and 20 weeks; then 12 weeks post-treatment
  Yale Brown Obsessive Compulsive Scale

SECONDARY OUTCOMES:
BDI-II Change | Prior to start; at 5 weeks, 10 weeks, 15 weeks, and 20 weeks; then 12 weeks post-treatment
  Beck Depression Inventory
QOLS Change | Prior to start; at 5 weeks, 10 weeks, 15 weeks, and 20 weeks; then 12 weeks post-treatment
  Quality Of Life Scale
Functions of Identity Scale Change | Prior to start; at 5 weeks, 10 weeks, 15 weeks, and 20 weeks; then 12 weeks post-treatment
  Examines aspects of identity
Social Connectedness Scale Change | Prior to start; at 5 weeks, 10 weeks, 15 weeks, and 20 weeks; then 12 weeks post-treatment
  Measure of sense of social connectedness

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams GR, Marshall SK. A developmental social psychology of identity: understanding the person-in-context. J Adolesc. 1996 Oct;19(5):429-42. doi: 10.1006/jado.1996.0041. PMID 9245296
- [Background] Cordier R, Milbourn B, Martin R, Buchanan A, Chung D, Speyer R. A systematic review evaluating the psychometric properties of measures of social inclusion. PLoS One. 2017 Jun 9;12(6):e0179109. doi: 10.1371/journal.pone.0179109. eCollection 2017. PMID 28598984
- [Background] Dembo JS. "The ickiness factor:" case study of an unconventional psychotherapeutic approach to pediatric OCD. Am J Psychother. 2014;68(1):57-79. doi: 10.1176/appi.psychotherapy.2014.68.1.57. PMID 24818457
- [Background] DeSocio JE. Accessing self-development through narrative approaches in child and adolescent psychotherapy. J Child Adolesc Psychiatr Nurs. 2005 Apr-Jun;18(2):53-61. doi: 10.1111/j.1744-6171.2005.00012.x. PMID 15966948
- [Background] Goncalves MM, Ribeiro AP, Silva JR, Mendes I, Sousa I. Narrative innovations predict symptom improvement: Studying innovative moments in narrative therapy of depression. Psychother Res. 2016 Jul;26(4):425-35. doi: 10.1080/10503307.2015.1035355. Epub 2015 May 13. PMID 25968420
- [Background] Goncalves MM, Stiles WB. Narrative and psychotherapy: introduction to the special section. Psychother Res. 2011 Jan;21(1):1-3. doi: 10.1080/10503307.2010.534510. No abstract available. PMID 21331976
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Richter PMA, Ramos RT. Obsessive-Compulsive Disorder. Continuum (Minneap Minn). 2018 Jun;24(3, BEHAVIORAL NEUROLOGY AND PSYCHIATRY):828-844. doi: 10.1212/CON.0000000000000603. PMID 29851880